CLINICAL TRIAL: NCT03945877
Title: Chronic Musculoskeletal Pain Experiences in Marginalized Populations: A Mixed Methods Study Protocol for Understanding the Impact of Geopolitical, Historical, and Societal Influences
Brief Title: Mixed Methods Study Protocol_Chronic Pain and Marginalized Populations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: High Point University (Other)
Collaborators: University of Otago (Other)
Responsible Party: Principal Investigator, Alicia Emerson, Assistant Professor, High Point University
Other Study IDs: HighPointU
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain; Marginalization, Social
MeSH Terms: conditions — Chronic Pain; Social Marginalization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- English-speaking Community Members: Survey respondents
  Interventions: Other: No interventions
- Spanish-speaking Community Members: Survey respondents
  Interventions: Other: No interventions
- Arabic-speaking Community Members: Survey respondents
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
A mixed-methods sequential explanatory design study. The first quantitative phase will be a multi-language survey that includes questions related to pain status, patient beliefs, pain interference/social support, and perspective on healthcare utilization. Latent class analysis (LCA) will be used to generate experience-based subgroups in CMP. The second qualitative phase will use focus group will elucidate, confirm, and more richly describe the findings from the first phase.

DETAILED DESCRIPTION:
Background: The global epidemic of chronic musculoskeletal pain (CMP) is an intractable issue adversely impacting gross domestic products and costing billions in lost productivity. The expansion of CMP occurs concurrently with historical global mass population movements. Geopolitical negative and racist rhetoric have arisen in response to increased immigration rates. CMP is an invisible disease decoupled from normal tissue healing and results from the complex interplay of biological and psychological processing. Different theoretical models of CMP development now include potential demographic and socio-cultural factors. CMP occurs disproportionately in populations at risk for marginalization, including women, non-Caucasians, immigrants, and people experiencing increased socioeconomic deprivation. The same marginalized populations also are at greater risk for limited access to healthcare and demonstrate worse functional limitations, outcomes, and quality of life. Aims: The primary aims are 1) to characterize self-reported features in people who have CMP and experience marginalization and 2) to interpret the pain experience for marginalised populations of people who have CMP. Methods: A mixed-methods sequential explanatory design study will be used. The first quantitative phase will be a multi-language survey that includes questions related to pain status, patient beliefs, pain interference/social support, and perspective on healthcare utilization. Latent class analysis (LCA) will be used to generate experience-based subgroups in CMP. Focus group will elucidate, confirm, and more richly describe the findings from the first phase. Discussion: Results from this study will be used to inform clinical conversations with patients who have CMP and experience marginalization. By increasing awareness of the potential influences on the clinical conversation, we hope to build opportunities to address inequities in CMP management.

ELIGIBILITY:
Inclusion Criteria:

* English, Spanish, and Arabic-speaking adults living in the Piedmont Triad, NC

Exclusion Criteria:

* declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: English-speaking adults who answer the phone and consent to participate. Spanish and Arabic-speaking adults who consent to participate in an in-person survey.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative: Community surveys | February 2017-September 2017
  Demographic data; Survey data
Qualitative: Focus groups | November 2018-December 2019
  Semi-structured interview data obtained from focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Emerson, PT, DPT, MS, Principal Investigator — High Point University and University of Otago
Locations (1):
- High Point University, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansfield KE, Sim J, Jordan JL, Jordan KP. A systematic review and meta-analysis of the prevalence of chronic widespread pain in the general population. Pain. 2016 Jan;157(1):55-64. doi: 10.1097/j.pain.0000000000000314. PMID 26270591
- [Background] Macfarlane GJ, Barnish MS, Jones GT. Persons with chronic widespread pain experience excess mortality: longitudinal results from UK Biobank and meta-analysis. Ann Rheum Dis. 2017 Nov;76(11):1815-1822. doi: 10.1136/annrheumdis-2017-211476. Epub 2017 Jul 21. PMID 28733474
- [Background] Fillingim RB, King CD, Ribeiro-Dasilva MC, Rahim-Williams B, Riley JL 3rd. Sex, gender, and pain: a review of recent clinical and experimental findings. J Pain. 2009 May;10(5):447-85. doi: 10.1016/j.jpain.2008.12.001. PMID 19411059
- [Background] Pedraza FI, Nichols VC, LeBron AMW. Cautious Citizenship: The Deterring Effect of Immigration Issue Salience on Health Care Use and Bureaucratic Interactions among Latino US Citizens. J Health Polit Policy Law. 2017 Oct;42(5):925-960. doi: 10.1215/03616878-3940486. Epub 2017 Jun 29. PMID 28663179
- [Background] Edwards RR, Moric M, Husfeldt B, Buvanendran A, Ivankovich O. Ethnic similarities and differences in the chronic pain experience: a comparison of african american, Hispanic, and white patients. Pain Med. 2005 Jan-Feb;6(1):88-98. doi: 10.1111/j.1526-4637.2005.05007.x. PMID 15669954
- [Background] Kim HJ, Yang GS, Greenspan JD, Downton KD, Griffith KA, Renn CL, Johantgen M, Dorsey SG. Racial and ethnic differences in experimental pain sensitivity: systematic review and meta-analysis. Pain. 2017 Feb;158(2):194-211. doi: 10.1097/j.pain.0000000000000731. PMID 27682208
- [Background] Green CR, Anderson KO, Baker TA, Campbell LC, Decker S, Fillingim RB, Kalauokalani DA, Lasch KE, Myers C, Tait RC, Todd KH, Vallerand AH. The unequal burden of pain: confronting racial and ethnic disparities in pain. Pain Med. 2003 Sep;4(3):277-94. doi: 10.1046/j.1526-4637.2003.03034.x. PMID 12974827
- [Background] Trost Z, Van Ryckeghem D, Scott W, Guck A, Vervoort T. The Effect of Perceived Injustice on Appraisals of Physical Activity: An Examination of the Mediating Role of Attention Bias to Pain in a Chronic Low Back Pain Sample. J Pain. 2016 Nov;17(11):1207-1216. doi: 10.1016/j.jpain.2016.08.001. Epub 2016 Aug 20. PMID 27555428
- [Background] Craig KD. Social communication model of pain. Pain. 2015 Jul;156(7):1198-1199. doi: 10.1097/j.pain.0000000000000185. No abstract available. PMID 26086113
- [Background] Harding G, Parsons S, Rahman A, Underwood M. "It struck me that they didn't understand pain": the specialist pain clinic experience of patients with chronic musculoskeletal pain. Arthritis Rheum. 2005 Oct 15;53(5):691-6. doi: 10.1002/art.21451. PMID 16208656
- [Background] Franklin ZC, Smith NC, Fowler NE. A qualitative investigation of factors that matter to individuals in the pain management process. Disabil Rehabil. 2016 Sep;38(19):1934-42. doi: 10.3109/09638288.2015.1107782. Epub 2016 Jan 4. PMID 26728636
- [Background] Burgess DJ, van Ryn M, Crowley-Matoka M, Malat J. Understanding the provider contribution to race/ethnicity disparities in pain treatment: insights from dual process models of stereotyping. Pain Med. 2006 Mar-Apr;7(2):119-34. doi: 10.1111/j.1526-4637.2006.00105.x. PMID 16634725
- [Background] Klonoff EA. Disparities in the provision of medical care: an outcome in search of an explanation. J Behav Med. 2009 Feb;32(1):48-63. doi: 10.1007/s10865-008-9192-1. Epub 2009 Jan 6. PMID 19127421